CLINICAL TRIAL: NCT02943083
Title: Promoting Mother-Baby Bonding Through a Relaxation Routine During Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: Johnson & Johnson (Industry)
Responsible Party: Principal Investigator, Elizabeth Werner, Assistant Professor of Behavioral Medicine (in Psychiatry) at CUMC, New York State Psychiatric Institute
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Supportive Care
Other Study IDs: 7244
Record Dates: First submitted 2016-10-13; First posted 2016-10-24 (Estimated); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Psychological Stress in Pregnancy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Coached Intervention (Experimental): Perform prenatal relaxation exercise in the lab with a coach and at home
  Interventions: Behavioral: Relaxation Exercise
- Home Intervention (Active Comparator): Only perform relaxation exercise at home
  Interventions: Behavioral: Relaxation Exercise
- Control Group (No Intervention): Never performs relaxation routine, attends prenatal assessment sessions
- Postpartum Only (No Intervention): Only attends visits postpartum, never receives prenatal assessments

INTERVENTIONS:
Behavioral: Relaxation Exercise — Groups receiving the intervention will be asked to engage in the relaxation protocol every day. Participants will be asked to continue practicing the relaxation protocol for the remainder of their pregnancy. Participants will be instructed to listen to the 7 minute guided muscle relaxation tape and engage in the 3 minute abdominal touch routine in the presence of the scent stick. Participants will be provided with a scent stick of their selected scent to take home. For the duration of the study, participants will be loaned standard headphones and an iPod Touch that contains only the guided progressive muscle relaxation audio recording to facilitate this at-home protocol.
  Arms: Coached Intervention; Home Intervention

SUMMARY:
The aims of this study are to determine if:

1. during pregnancy, a progressive muscle relaxation and abdominal touch ritual involving a pleasing scent (i.e. a "relaxation ritual") can, acutely, reduce maternal stress and affect the fetus (in terms of movement, changes in heart rate and heart rate variability);
2. a progressive muscle relaxation and abdominal touch ritual involving a pleasing scent (i.e. a "relaxation ritual") during pregnancy can have an effect on mitochondria functioning in the placenta through reducing maternal stress during pregnancy (based on our recent findings (Monk et al, 2016));
3. the scent will come to function as a conditioned stimulus such that exposure to the scent postpartum will induce greater maternal relaxation, which will have an effect on the mother-infant interaction and infant physiology;
4. prenatal maternal exposure to scent combined with abdominal touch will lead to mothers' increased likelihood of utilizing infant massage with a lotion of the same scent postpartum;
5. the prenatal ritual and the increased likelihood of engaging in infant massage will lead to a maternal perception of greater mother-infant bonding, attachment and parenting efficacy, and improved maternal mood;
6. the prenatal ritual and the increased likelihood of engaging in infant massage will lead to improved performance on the conjugate reinforcement paradigm conditioning task administered to infants at 4 months of age

DETAILED DESCRIPTION:
Some women will randomly be assigned to perform the prenatal relaxation ritual both in our lab and at home (Coached Intervention (CI)); some to make prenatal visits to the lab but perform the prenatal relaxation ritual at home only (Home Intervention (HI)); and some to make prenatal visits to the lab but never to perform the prenatal relaxation ritual (Control Group (CG)). In addition, a fourth group of participants will participate in postpartum sessions only (Postpartum Only Group (PO)); the only prenatal experience these participants will have in the laboratory will be the informed consent session. Participants in all four groups (CI, HI, CG, PO) will participate in an informed consent and demographic information session prenatally, during which demographic information and medical history will be collected. At the informed consent and demographic information session, women who participate in prenatal sessions (those in CI, HI and CG) will smell three scent sticks and select their favorite scent. Women in the relaxation ritual groups (those in CI and HI) will utilize the scent in the relaxation ritual during pregnancy. Women in the CG will not be exposed to the scent again until the postpartum period (as detailed in the description of postpartum sessions, below). After the informed consent session, women who participate in prenatal sessions (those in CI, HI and CG) will come into the lab three times for the prenatal sessions, during which participants will be administered questionnaires about background information, moods and stress; collect hair samples for analysis of the stress hormone cortisol; collect blood and saliva samples for analysis of the hormone oxytocin, which plays a role in social interaction, bonding and lactation; and conduct fetal sessions to simultaneously collect maternal and fetal heart rate, as well as maternal blood pressure and respiration and fetal movement. Women in the group that performs the relaxation ritual in the lab (CI) will perform the ritual during the fetal sessions; this will allow assessment of any acute affects of the ritual on mom and fetus. In order to assess if the relaxation ritual during pregnancy can have an effect on mitochondria functioning in the placenta, placentas will be collected from all participants post-delivery and stored for future analyses.

All women will participate in a postpartum session in the hospital within 36 hours of birth. At this session, women in the PO group will have the opportunity to smell the same scent sticks that the other groups smelled prenatally, and select a favorite scent. All women will be given a scented lotion, matching the scent participants were exposed to either prenatally (CI and HI), that participants chose prenatally for postpartum use (CG) or that participants had just selected postpartum (PO). All women will apply the scented lotion and pick up their babies at this session. During this holding period, the investigators will monitor mother and baby heart rate and respiration and baby brain activity via EEG to assess maternal and infant relaxation. Afterwards, all women will be given information on how to use the lotion to give a gentle infant massage.

All dyads will also participate in a 6-week taped diapering and lotion session; the tape will be coded for quality of mother-infant interaction to assess dyadic affect and bonding. Participants will also participate in a session 4-months postpartum where infants engage in a neurocognitive test that assesses memory through a kicking task (conjugate reinforcement paradigm conditioning task). Women will answer questionnaires about their moods, how participants feel about their babies and their babies' daily routines at both of these sessions.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant women between 18-45 years old,Self-report
2. Not smoking during pregnancy,Self-report
3. Healthy pregnancy,Self-report
4. 26 weeks ± 3 weeks gestation by time of enrollment,Self-report
5. Delivering baby at CUMC- CHONY or Allen Pavilion,Self-report
6. Receiving prenatal care,Self-report

Exclusion Criteria:

1. Multi-fetal pregnancy, Selfreport
2. Taking medications that affect the cardiovascular system (α blockers, β blockers, corticosteroids, chronic-use asthma medications (e.g. beta2-adrenoceptor agonists), Selfreport
3. Drinking alcohol or using recreational drugs during pregnancy, Selfreport
4. Premature birth (before 37.5 weeks gestation)*, Medical record

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 106 (Estimated)
Dates: Start 2016-10; Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Mother-Infant Bonding assessed by Postpartum Bonding Questionnaire | 6 weeks to 4 months postpartum
  Improved level of mother-infant bonding as assessed by Postpartum Bonding Questionnaire

SECONDARY OUTCOMES:
Change in Maternal Stress Level during Pregnancy as assessed by Perceived Stress Scale | Change over time from 24 weeks gestation to 36 weeks gestation
  Reduction in stress as operationalized through Perceived Stress Scale

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Monk, Ph.D., Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No